CLINICAL TRIAL: NCT01105962
Title: Multicenter Observational Study of Hyperbaric Oxygen Therapy (HBOT) in Chronic Traumatic Brain Injury (TBI)/Post-Concussion Syndrome (PCS) and/or TBI/Post-Traumatic Stress Disorder (PTSD)
Brief Title: Hyperbaric Oxygen Therapy in Chronic Traumatic Brain Injury or Post-Traumatic Stress Disorder
Acronym: NBIRR-1
Status: Terminated | Type: Observational
Why Stopped: new regulatory requirements will require funding for restart as a new study
Sponsor: International Hyperbaric Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NBIRR-01
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Traumatic Brain Injury; Post-traumatic Stress Disorder
Keywords: traumatic; brain; injury; post-traumatic; stress; hyperbaric; oxygen; HBOT; TBI; PTSD
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an observational research study whose purposes are to see:

1. if 40 Hyperbaric Oxygen Therapy sessions at 1.5 atmospheres (HBOT 1.5) or more (60, or 80 HBOT's) help, worsen, or have no effect on subjects with chronic TBI/PCS (Traumatic Brain Injury/Post-Concussion Syndrome) and/or PTSD (Post-Traumatic Stress Disorder).
2. if improvements or worsening of symptoms can be recorded with computerized and written tests for memory and thinking, and with questionnaires about the subject's quality of life and health.
3. determine the long-term outcome of the treatment.
4. confirm, in large numbers of study participants at multiple sites nationwide, the strong positive results obtained in pilot studies

ELIGIBILITY:
Inclusion Criteria:

1. Any 18-65 year-old patient with mild-moderate TBI or PTSD. (If a military injury, subject may be active duty or a veteran. If active duty, participants will have to voluntarily contact NBIRR.)
2. Have demonstrated a >20% decrement (compared to pre-deployment baseline) in ANAM composite score or specific sub-score with regard to "simple reaction time" and/or "procedural reaction time".
3. Have a diagnosis of TBI, chronic TBI/PCS or TBI/PCS/PTSD or PTSD made by a military (military etiology of blast injury) or civilian specialist.
4. Negative pregnancy test in females.
5. Less than 90% on the Percent Back to Normal Rating Scale. (If patient is considered 100% normal before TBI, patient should be less than 90% normal for entry into the study).

Exclusion Criteria:

1. Pulmonary disease that precludes HBOT (e.g., asthma unresponsive to medication, bullous emphysema).
2. Unstable medical conditions that are contraindicated in HBOT (e.g. severe congestive heart failure or heart failure requiring hospital emergency evaluation or admission in the previous year).
3. Severe confinement anxiety (claustrophobia; e.g., patients who require anesthesia conscious sedation for MRI or who cannot go in elevators).
4. Pregnancy.
5. Other pre-TBI neurological diagnoses.(seizure disorders, multiple sclerosis, Parkinson's, Lyme, etc.)
6. Participation in another experimental trial with active intervention.
7. High probability of inability to complete the experimental protocol (e.g. terminal condition).
8. Past or current history of mental retardation unless diagnosed post TBI (baseline IQ ≤ 70).
9. Pre- or post-TBI history of systemic illness with impact on central nervous system. (Principal Investigator in consultation with study sponsor Medical Officer will make the ultimate decision).
10. Any pre-existing chronic infection not related to battlefield injuries or government service.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One thousand subjects will be recruited. Subjects will be 18-65 years old and have been diagnosed with mild or moderate (but not severe) TBI or TBI/PTSD or PTSD by either the military (any etiology) or civilian neurologists or neuropsychologists. This diagnosis will especially include war veterans who have had a significant decrease in their neuropsychological test scores.
  There will be no gender restriction. However, it is anticipated that the cohort will consist mostly of males, due to the nature of the injury. There will be no race or ethnicity restriction.
  All subjects will be legally capable of consenting. No subjects who need 3rd party consent will be enrolled in the NBIRR study.
  Military - Unless specifically approved by a military site IRB, active duty participants will have to voluntarily contact NBIRR participating sites or respond to a recruitment outreach outside of the command.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Function | 2-6mo then every 6 months for 2yrs

CONTACTS AND LOCATIONS:
Overall Officials: B Robert Mozayeni, MD, Study Director — International Hyperbaric Medical Foundation
Locations (10):
- United States (10):
  - San Francisco Institute for Hyperbaric Medicine, San Francisco, California
  - Rocky Mountain Hyperbaric Institute, Boulder, Colorado
  - Hyperbaric Services of the Palm Beaches, Delray Beach, Florida
  - Hyperbaric Medicine Inc. of Florida, Fort Walton Beach, Florida
  - Idaho Wound Care & Hyperbaric Medicine, Pocatello, Idaho
  - Lifeforce Therapies, Plymouth, Minnesota
  - Hyperbaric Institute of Nevada and Clinical Neurology Specialists, Henderson, Nevada
  - Alliance Community Hospital Wound Care and Hyperbaric Department, Alliance, Ohio
  - HBOT NOVA - Hyperbaric Oxygen Therapy of Northern Virginia, Reston, Virginia
  - Fox Valley Wellness Center, Fond du Lac, Wisconsin

REFERENCES:
- See also: National Brain Injury Rescue and Rehabilitation Project — http://www.nbirr.org